CLINICAL TRIAL: NCT01301950
Title: Comparison of Surgical Time and Efficiency of Total Knee Arthroplasty Using TruMatch® Personalized Solutions Compared to Conventional Total Knee Arthroplasty
Brief Title: Comparison of Surgical Time and Efficiency of Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08004
Record Dates: First submitted 2010-12-02; First posted 2011-02-23 (Estimated); Results first posted 2014-09-05 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Osteoarthritis, Knee
Keywords: Arthroplasties, Knee Replacement; Arthroplasties, Replacement, Knee; Arthroplasty, Knee Replacement; Knee Replacement Arthroplasties; Knee Replacement Arthroplasty; Knee Replacement, Total; Replacement Arthroplasties, Knee; Replacement Arthroplasty, Knee; Replacement, Total Knee; Total Knee Replacement
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TruMatch® Personalized Solutions (Active Comparator): Cruciate Retaining and Posterior Stabilized Fixed-Bearing or Rotating Platform Total Knee Arthroplasty (PFC Sigma System) implanted using TruMatch® Personalized Solutions (Custom Patient Instrumentation)
  Interventions: Other: Custom Patient Instrumentation
- Conventional Total Knee Replacement (Active Comparator): Cruciate Retaining and Posterior Stabilized Fixed-Bearing or Rotating Platform Total Knee Arthroplasty (PFC Sigma System) implanted using conventional instruments
  Interventions: Other: Conventional Instruments

INTERVENTIONS:
Other: Custom Patient Instrumentation — TruMatch® Personalized Solutions is the brand name of DePuy Orthopaedics, Inc. custom patient instrumentation (CPI). TruMatch™ is a pair of custom-made cutting blocks that allow distal femoral and proximal tibial cuts to be made according to a predefined surgical plan. The inner surface of the femoral block is manufactured to match the geometry of the patient's distal femur. The inner surface of the tibial block is manufactured to match the patient's proximal tibia. The geometric data is obtained from a CT scan and a preoperative plan approved by the surgeon
  Other Names: TruMatch® Personalized Solutions
  Arms: TruMatch® Personalized Solutions
Other: Conventional Instruments — Total Knee Arthroplasty implanted using conventional instruments (non-CPI) and surgical technique.
  Arms: Conventional Total Knee Replacement

SUMMARY:
This study is designed to compare the surgical efficiency of TruMatch® Personalized Solutions surgical technique compared to conventional surgical technique. Specifically, the purpose of this study is to collect time data to enhance the existing economic model.

DETAILED DESCRIPTION:
The study is designed as a prospective, multi-center, controlled, non-randomized, clinical investigation to compare the efficiency of TruMatch® Personalized Solutions surgical technique compared to conventional surgical technique.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female and between the ages of 18 and 80 years old, inclusive.
* Subject requires a primary total knee replacement and is considered by the Investigator to be suitable for the specific knee prosthesis identified in the protocol.
* Subject has given voluntary, written informed consent to participate in this clinical investigation and has authorized the transfer of his/her information to DePuy
* Subject, in the opinion of the Clinical Investigator, is able to understand this clinical investigation, and co-operate with investigational procedures.
* Subject, who, in the opinion of the Clinical Investigator, are suitable for implantation using TruMatch™ instrumentation. For example, no femoral nails/bone plates that extend into the knee, ie. within 8cm of joint line; no metal device that could cause CT scatter about the knee and no deformities greater than 15 degrees of fixed varus, valgus, or flexion contracture are consistent with TruMatch™ instrumentation.

Exclusion Criteria:

* The Subject is a woman who is pregnant or lactating.
* The Subject has participated in a clinical investigation with an investigational product in the last 3 months.
* The Subject is currently involved in any personal injury litigation, medical-legal or worker's compensations claims.
* The Subject has previously had a prosthetic knee replacement device (any type) of the affected knee.
* The Subject requires simultaneous bilateral total knee replacements.
* The Subject had a contralateral TKA and that knee was previously entered in the study.
* Subject in whom the surgeon intends to implant a knee prosthesis that is not in the PFC Sigma primary knee system.
* Subject who has inflammatory arthritis.
* Subject who has a Body Mass Index (BMI) of ≥ 40. (Please see Table 2-1: Definition of Terms, for BMI definition and calculation formulas).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2013-08-01 (Actual); Study Completion 2013-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Painter, Principal Investigator — Pinnacle Orthopaedics
Locations (3):
- United States (3):
  - Center for Hip and Knee Surgery, Mooresville, Indiana
  - Pinnacle Orthopaedics, Bartlesville, Oklahoma
  - Commonwealth Orthopaedics, Reston, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- TruMatch® Personalized Solutions: Cruciate Retaining and Posterior Stabilized Fixed-Bearing or Rotating Platform Total Knee Arthroplasty (P.F.C. Sigma System) implanted using TruMatch® Personalized Solutions. Instrument: TruMatch® Personalized Solutions is the brand name of DePuy Orthopaedics, Inc. custom patient instrumentation. TruMatch® is a pair of custom-made cutting blocks that allow distal femoral and proximal tibial cuts to be made according to a predefined surgical plan. The inner surface of the femoral block is manufactured to match the geometry of the patients' distal femur. The inner surface of the tibial block is manufactured to match the patient's proximal tibia. The geometric data is obtained from a CT scan and a preoperative plan approved by the surgeon.
Period: Overall Study
Arm/Group | Conventional Total Knee Replacement | TruMatch® Personalized Solutions
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Surgery was cancelled by patient | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects who were consented prior to surgery were included in the analysis of baseline characteristics.
Groups:
- TruMatch® Personalized Solutions: Cruciate Retaining and Posterior Stabilized Fixed-Bearing or Rotating Platform Total Knee Arthroplasty (PFC Sigma System) implanted using TruMatch® Personalized Solutions Instrument: TruMatch® Personalized Solutions is the brand name of DePuy Orthopaedics, Inc. custom patient instrumentation. TruMatch® is a pair of custom-made cutting blocks that allow distal femoral and proximal tibial cuts to be made according to a predefined surgical plan. The inner surface of the femoral block is manufactured to match the geometry of the patient's distal femur. The inner surface of the tibial block is manufactured to match the patient's proximal tibia. The geometric data is obtained from a CT scan and a preoperative plan approved by the surgeon
- Total: Total of all reporting groups
Arm/Group | TruMatch® Personalized Solutions | Conventional Total Knee Replacement | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (12.9) | 62.7 (9.1) | 62.8 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 9 | 4 | 13
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Surgical Procedure Time to Compare Skin-to-Skin Time for Conventional Versus TruMatch® Primary Total Knee Replacements
Description: Skin-to skin time for conventional versus TruMatch® primary total knee replacements (recorded by Investigator on Operative case report forms).
Time Frame: Intraoperative (Time from first incision to first stitch)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Conventional Total Knee Replacement | TruMatch® Personalized Solutions
Number analyzed (Participants) | 15 | 14
minutes | 65.8 (12.3) | 67.3 (20.6)
Statistical Analysis 1: Comparison: Conventional Total Knee Replacement vs TruMatch® Personalized Solutions; The null hypothesis was no difference in skin-to-skin time. The alternative hypothesis was that the TruMatch group time was less than the conventional group. Statistical power was anticipated to be 86% with 40 enrolled subjects based upon a Cohen's D effect size of 1. The Sponsor had difficulty identifying and recruiting sites suitable for participation. The statistically required sample size (N=40) was therefore not obtained, causing the group comparison to be statistically underpowered; Test type: Superiority or Other; p = 0.54, ANOVA

2. Secondary Outcome: Operating Room Setup - Operating Room Cleaned up From Previous Case to Surgical Draping Complete
Description: Operating Room setup time for conventional versus TruMatch® primary total knee replacements as recorded by video time analysis [minutes]
Time Frame: Intraoperative (Operating Room cleaned up from previous case to surgical draping complete)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Conventional Total Knee Replacement | TruMatch® Personalized Solutions
Number analyzed (Participants) | 15 | 14
minutes | 28.9 (15.0) | 28.8 (14.4)

3. Secondary Outcome: Turnover Time (Time to Clean Operating Room After Surgery is Completed)
Description: Turnover Time for conventional versus TruMatch® primary total knee replacements as recorded by video time analysis [minutes].
Time Frame: Intraoperative (Time to clean Operating Room after surgery is completed)
Population: 1 site (9 subjects) was excluded from Turnover Time analysis as this substep could not be accurately assessed due to unexpected difficulties during video collection.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Conventional Total Knee Replacement | TruMatch® Personalized Solutions
Number analyzed (Participants) | 10 | 10
minutes | 10.1 (4.8) | 11.4 (2.8)

4. Secondary Outcome: Costs Associated With Conventional Versus TruMatch® Total Knee Arthroplasty Surgical Procedures
Description: Compare costs associated with surgery using conventional surgical technique versus TruMatch® primary total knee replacements .
Time Frame: Intraoperative (Total duration of procedure)
Population: No cost data were collected, resulting in a sample size of 0.
Arm/Group | Conventional Total Knee Replacement | TruMatch® Personalized Solutions
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: To Compare the Differences in Operating Room Efficiency as a Function of Institution Type and Geographical Location
Time Frame: Intraoperative
Population: No operating room efficiency data was analyzed as a function of geography and institution, resulting in a sample size of 0.
Arm/Group | Conventional Total Knee Replacement | TruMatch® Personalized Solutions
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Intraoperative
Groups:
- TruMatch™ Personalized Solutions: Cruciate Retaining and Posterior Stabilized Fixed-Bearing or Rotating Platform Total Knee Arthroplasty (PFC Sigma System) implanted using TruMatch™ Personalized Solutions Instrument: TruMatch™ Personalized Solutions is the brand name of DePuy Orthopaedics, Inc. custom patient instrumentation. TruMatch™ is a pair of custom-made cutting blocks that allow distal femoral and proximal tibial cuts to be made according to a predefined surgical plan. The inner surface of the femoral block is manufactured to match the geometry of the patient's distal femur. The inner surface of the tibial block is manufactured to match the patient's proximal tibia. The geometric data is obtained from a CT scan and a preoperative plan approved by the surgeon
Arm/Group | TruMatch™ Personalized Solutions | Conventional Total Knee Replacement
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 0/14 | 0/15

LIMITATIONS AND CAVEATS:
A statistically powered sample size was not obtained; Two secondary objectives (compare costs & compare differences in OR efficiency as a function of institution type & geographic location) could not be assessed as originally intended by the protocol

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less